CLINICAL TRIAL: NCT00869362
Title: Effect of Inpatient Diabetes Management on Outpatient Glycemic Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Deborah Wexler, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008P-001439; K23DK080228 (NIH)
Record Dates: First submitted 2009-03-25; First posted 2009-03-26 (Estimated); Results first posted 2012-11-02 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetes Management Team (Experimental): Evaluation and management by diabetes management team
  Interventions: Other: Diabetes management team
- Control (No Intervention): Patients receive usual care for diabetes

INTERVENTIONS:
Other: Diabetes management team — MD evaluation followed by NP education and and medication titration
  Arms: Diabetes Management Team

SUMMARY:
The hypothesis of this study is that using hospital admission to identify patients with poorly controlled diabetes (hemoglobin A1c levels >8%), and intervening during the hospitalization with targeted inpatient diabetes management will improve glycemic control at 3 and 12 months, with inpatient glycemic control, quality of life, and diabetes self-efficacy serving as secondary endpoints.

DETAILED DESCRIPTION:
The study is a randomized, controlled trial of targeted inpatient diabetes management versus usual care in 70 general medical and surgical inpatients over age 18 with type 2 diabetes and hemoglobin A1c levels greater than 8% who are followed in Partners-affiliated primary care practices. In addition, we will enroll a prospective chart review cohort matched for age, sex, and HbA1c level whose course we will follow for one year after discharge to determine the patter of glycemia among patients who are not enrolled in a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Known diagnosis of type 2 diabetes by history with outpatient prescription of oral hypoglycemic medication or insulin
* Hemoglobin A1c > 8.0% within the prior 12 months, or if not known, fasting blood glucose greater than 200 mg/dl on sliding scale regular insulin.
* Partners-affiliated primary care physician

Exclusion Criteria:

* Screening HbA1c returns less than 8%.
* Diabetic ketoacidosis (DKA) as a primary reason for admission (admission blood glucose > 250 mg/dl with arterial pH < 7.30 or serum bicarbonate level < 15 mg/dl), or development of DKA during admission.
* Hyperosmolar hyperglycemic syndrome as a primary reason for admission (admission blood glucose > 400 mg/dl and plasma osmolality > 315 mOsm/kg.
* Pregnancy, ruled out by urine HCG test at screening after consent is obtained in all women who continue to have menstrual cycles.
* Anemia with hemoglobin < 9 g/dl, recent blood transfusion, or need for blood transfusion (interferes with interpretation of hemoglobin A1c assay)
* End stage liver disease with prothrombin time > 15 seconds and albumin <3 mg/dl
* End stage renal disease: Stage IV (glomerular filtration rate <30 mg/dl) or V chronic kidney disease
* Treatment with corticosteroids
* ICU transfer
* Inability to self-administer insulin
* Hypoglycemia unawareness: patient lacks sensation of common signs of blood glucose < 60 mg/dl (tachycardia, diaphoresis, hunger, confusion, fatigue).
* Projected survival < 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2009-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah J Wexler, MD, MSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Wexler DJ, Beauharnais CC, Regan S, Nathan DM, Cagliero E, Larkin ME. Impact of inpatient diabetes management, education, and improved discharge transition on glycemic control 12 months after discharge. Diabetes Res Clin Pract. 2012 Nov;98(2):249-56. doi: 10.1016/j.diabres.2012.09.016. Epub 2012 Oct 1. PMID 23036785

RESULTS

PARTICIPANT FLOW:
Recruitment Details: April, 2009 to May 2010, recruited from inpatient medical and surgical general care (non-ICU) inpatient units
Groups:
- Diabetes Management Team: Evaluation and management by diabetes management team including physician and nurse practitioner CDE. Physician performed diabetes medication initiation and/or titration and nurse performed CDE focusing on Diabetes Survival Skills.
Period: Overall Study
Arm/Group | Diabetes Management Team | Control
Started | 15 | 16
Completed | 14 | 11
Not Completed | 1 | 5
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Diabetes Management Team | Control | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 11 | 21
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.2 (11.3) | 52.9 (13.7) | 55 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  United States | 15 | 16 | 31

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c
Description: Change in glycemic control measured by HbA1c change baseline to 6 months
Time Frame: 6 months from discharge
Measure: Mean (Standard Deviation); unit: HbA1c, %
Groups:
- Diabetes Management Team: Evaluation and management by diabetes management team (physician, nurse practitioner CDE) with physician-initiation and titration of diabetes medication and nurse CDE education on Diabetes Survival Skills.
Arm/Group | Diabetes Management Team | Control
Number analyzed (Participants) | 15 | 16
HbA1c, % | -1.3 (2.3) | -0.4 (1.1)

2. Secondary Outcome: Average Intervention Effect Over 12 Months After Hospital Discharge
Time Frame: 12 months from discharge
Measure: Mean (Standard Error); unit: HbA1c, %
Arm/Group | Diabetes Management Team | Control
Number analyzed (Participants) | 15 | 16
HbA1c, % | -0.6 (0.5) | -0.6 (0.5)

ADVERSE EVENTS:
Arm/Group | Diabetes Management Team | Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 2/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetes Management Team (N=15) | Control (N=16)
Death (Cardiac disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No